CLINICAL TRIAL: NCT07076537
Title: A Randomized Placebo Controlled Clinical Study on the Effects of a Dietary Supplement on Stress, Anxiety, Mood and Sleep in a Pediatric Population
Brief Title: A Clinical Study on the Effects of a Dietary Supplement on Stress, Anxiety, Mood and Sleep in a Pediatric Population
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Olly, PBC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: ULOLLYKC2
Record Dates: First submitted 2025-06-12; First posted 2025-07-22 (Actual); Last update posted 2025-07-22 (Actual); Status verified 2025-07

CONDITIONS: Healthy
MeSH Terms: interventions — Dietary Supplements

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Oral dietary supplement. Instructions: Take 2 gummies per day as needed. Chew thoroughly before swallowing. Ideally, take in the morning at the same time between 8:00 a.m. and 11:00 a.m.
  Interventions: Dietary Supplement: Placebo
- Dietary Supplement with actives (Active Comparator): Oral dietary supplement. Instructions: Take 2 gummies per day as needed. Chew thoroughly before swallowing. Ideally, take in the morning at the same time between 8:00 a.m. and 11:00 a.m.
  Interventions: Dietary Supplement: Dietary Supplement with actives

INTERVENTIONS:
Dietary Supplement: Placebo — Placebo
  Arms: Placebo
Dietary Supplement: Dietary Supplement with actives — Dietary Supplement containing magnesium, L-theanine and lemon balm extract
  Arms: Dietary Supplement with actives

SUMMARY:
The study will be a randomized, placebo control clinical study to assess the the efficacy for improvement of mood/stress and anxiety compared to placebo through validated survey questionnaire. The target population of this study is 5 to 14 years old. Participants will be asked to take questionnaires to collect baseline at the beginning of the study. The questionnaires are: Perceived Stress Scale for children (PSS-ch), The Positive Affect and Negative Affect Schedule-Child Form-children (PANAS-children) and the Children's Sleep Habits Questionnaire (CSHQ). The interventional treatment will be for a total of 4 weeks (28 days). Participants will be asked to take the questionnaires at the end of the 28 days. The subjects will attend two appointments in the clinic throughout the duration of the study.

DETAILED DESCRIPTION:
For these scale, here are some more details:

The PSS-C:

Scoring range: Each item is scored from 0 (Never) to 4 (Very Often), giving a total score range from 0 to 56.

Interpretation: Higher scores indicate higher perceived stress, meaning a worse outcome.

The PANAS-C:

Scoring range: Each item is rated on a scale from 1 (Very slightly or not at all) to 5 (Extremely), resulting in:

* Positive Affect (PA): 15 to 75
* Negative Affect (NA): 15 to 75

Interpretation:

Higher PA scores indicate more positive emotions (a better outcome) Higher NA scores indicate more negative emotions (a worse outcome)

The CSHQ Scoring range: Each item is scored as follows - 1 (Rarely), 2 (Sometimes), 3 (Usually). This gives a total score range from 33 to 99.

Interpretation: Higher scores suggest more disturbed or problematic sleep patterns, meaning a worse outcome.

ELIGIBILITY:
Inclusion Criteria:

1. Willingness to actively participate in the study and to come to the scheduled visits.
2. Healthy (Healthy as determined by medical history as assessed by Qualified Investigator ) female and male subjects in good health between 5 to 14 years old.
3. Enrolled in and currently attending school at baseline and for the duration of the study period.
4. Agreement to adhere to the procedures and requirements of the study and to report to the institute on the day(s) and at the time(s) scheduled for the assessments.
5. Ability to give consent (assent) for participation in the study

Exclusion Criteria:

1. Diagnosed with any mental health condition including chronic stress, GAD, impaired cerebral function, mood disorders, ADHD or similar conditions
2. Currently taking any prescription medications or dietary supplements for sleep, anxiety, depression or ADHD
3. Liver dysfunction
4. Use of sleep aides including dietary supplements over the past 7 days
5. History of reaction to the category of product tested
6. Other diseases or medications that might directly interfere in the study or put the subject's health under risk.
7. Participants having an acute or chronic disease or medical condition could put him/her at risk in the opinion of the Principal Investigator or compromise study outcomes.
8. Typical uncontrolled chronic or serious disease and/or conditions which would prevent participation in any clinical trials such as cancer, AIDs, diabetes, renal- impairment, mental illness, drug/alcohol addiction.
9. Subjects with a history of cancer within the past 5 years.
10. Subjects with any planned surgeries and/or invasive medical procedures during the study.
11. Individuals unable to communicate or cooperate with the principal investigator due to language
12. Employees (and children of employees) of TKL and/or product brand owner or manufacturer.

Ages: 5 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 80 (Estimated)
Dates: Start 2025-07-15 (Estimated); Primary Completion 2025-08-15 (Estimated); Study Completion 2025-09-02 (Estimated)

PRIMARY OUTCOMES:
To assess the efficacy for improvement of feelings of stress compared to placebo through validated survey questionnaire. | from enrollment to end of study at Week 4
  PSS-children will be administered before the intervention to establish baseline, 40 min after taking the initial dose and after taking the product for 28 days consecutively. Scores will be analyzed to assess changes in improvement in stress levels across the active and placebo arms. Data will be compared between the active supplement and placebo groups.
  More details on the scales
  The PSS-C: (perceived stress scale -children form) Scoring range: Each item is scored from 0 (Never) to 4 (Very Often), giving a total score range from 0 to 56.
  Interpretation: Higher scores indicate higher perceived stress, meaning a worse outcome.

SECONDARY OUTCOMES:
To assess the efficacy for improvement of feelings of positive and negative mood, and anxiety compared to placebo through validated survey questionnaire. | from enrollment to end of study at Week 4
  PANAS-children questionnaire will be administered before the intervention, to establish baseline, 40 min after initial dose and after taking the product for 28 days consecutively. Scores will be analyzed to assess changes in improvement of positive and negative mood across the active and placebo arms. Data will be compared between the active supplement and placebo groups.
  More details on scale:
  The PANAS-C: (positive and negative affect scale-children form)
  Scoring range: Each item is rated on a scale from 1 (Very slightly or not at all) to 5 (Extremely), resulting in:
  * Positive Affect (PA): 15 to 75
  * Negative Affect (NA): 15 to 75
  Interpretation:
  Higher PA scores indicate more positive emotions (a better outcome) Higher NA scores indicate more negative emotions (a worse outcome)
To assess the efficacy for improvement of sleep quality compared to placebo through validated survey questionnaire. | from enrollment to end of study at Week 4
  CSHQ questionnaire will be administered before the intervention, to establish baseline, and after taking the product for 28 days consecutively. Scores will be analyzed to assess changes in improvement sleep quality across the active and placebo arms. Data will be compared between the active supplement and placebo groups.
  More details on scale:
  The CSHQ (children sleep habits questionnaire) Scoring range: Each item is scored as follows - 1 (Rarely), 2 (Sometimes), 3 (Usually). This gives a total score range from 33 to 99.
  Interpretation: Higher scores suggest more disturbed or problematic sleep patterns, meaning a worse outcome.

CONTACTS AND LOCATIONS:
Locations (1):
- TKL Research, Fair Lawn, New Jersey, United States